CLINICAL TRIAL: NCT03862261
Title: Integrating Pediatric TB Services Into Child Healthcare Services in Africa. A Cluster-randomized Stepped-wedge Trial
Brief Title: Integrating Pediatric TB Services Into Child Healthcare Services in Africa
Acronym: INPUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: UNITAID (Other); University of Sheffield (Other); Kenya Ministry of Health (Other Government); Cameroon Ministry of Public Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: EG0214
Record Dates: First submitted 2019-02-12; First posted 2019-03-05 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Tuberculosis; Children, Only; Diagnosis; Delivery of Health Care
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Intervention Model Description: Cluster-randomized stepped-wedge model, where intervention will be randomly allocated to the different study sites at different time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-Care (No Intervention): Pediatric TB services based on current routine approach (national standard of care)
- Intervention (Experimental): Integrated pediatric TB services
  Interventions: Other: Integrated pediatric TB services

INTERVENTIONS:
Other: Integrated pediatric TB services — pediatric TB services will be integrated into key child healthcare services: maternal neonatal and child health (MNCH) services, under-5 clinic, pediatric outpatient services, nutrition services, pediatric antiretroviral therapy (ART) services and primary health care:
  * Integration of the screening into all the child health care services with introduction of a specific case detection tool and updated presumptive TB register.
  * Improvement of diagnosis capacities and their integration in all levels of care and all services.
  Arms: Intervention

SUMMARY:
Under-diagnosis of TB in children is a critical gap to address. The INPUT study is a multinational stepped-wedge cluster-randomized intervention study aiming to assess the effect of integrating TB services into child healthcare services on TB diagnosis capacities in children under 5 years of age.

DETAILED DESCRIPTION:
Study clusters (district-level hospitals and their health centers) will start under standard-of-care and transition to the intervention at randomly assigned time points.

In this study two strategies will be compared: i) The standard of care, offering pediatric TB services based on current routine approach; ii) The intervention, with pediatric TB services integrated into child healthcare services.

The primary objective will be to assess the effect of the intervention compared to standard of care on the proportion of TB cases diagnosed among children <5 years old (that is the number of children who are clinically or bacteriologically diagnosed with TB over the total number of children attending the child healthcare services). Secondary objectives are detailed in the protocol.

Study sites will include six hospital in each participating country (Cameroon and Kenya) along with selected attached health centers.

The study population will be children aged less than five years of age with a presumptive diagnosis of TB.

Study enrollment will start in March 2019, last enrollments until July 2020 and follow up will be completed by August 2021.

ELIGIBILITY:
Inclusion Criteria:

* Children < 5 years old.
* TB diagnosis investigations initiated.
* Other infectious diseases are not suspected or have already been ruled out.
* Commitment to take treatment in the clinic of enrolment or another INPUT study site.
* Parental/caregiver consent for the child to participate in the study.

Exclusion Criteria:

* Children who are TB contacts but without symptoms or signs of active TB

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1715 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of children diagnosed with active TB | up to two months
  Number of pediatric TB cases diagnosed (bacteriologically confirmed and/or clinically diagnosed) over the number of children attending the child healthcare services during the study period.

SECONDARY OUTCOMES:
Proportion of children screened for TB | one month
  Number of children screened for TB over the number of children attending the child healthcare services during the study period
Proportion of screened children who have a sample collected | up to three months
  Proportion of children who have a sample collected for microbiologic diagnosis among those screened positive for TB (i.e. presumptive TB cases)
Proportion of children diagnosed with TB among presumptive TB cases | up to two months
  Proportion of children diagnosed with TB (bacteriologically or clinically) among presumptive TB cases, overall and disaggregated by HIV status and nutrition status
Time from screening to clinical or bacteriologic diagnosis | up to three months
  For children finally diagnosed with TB, time elapsed from presumptive to confirmed TB case
Time from diagnosis to treatment initiation | up to three months
  For children diagnosed with TB, time elapsed to initiate treatment after active TB is confirmed
Proportion of cases with a bacteriologically confirmed diagnosis | up to three months
  Proportion of cases with a bacteriologically confirmed diagnosis among children diagnosed with TB
Proportion of children who initiate TB treatment among those diagnosed | up to two months
  Proportion of children who initiate TB treatment among those diagnosed will give treatment coverage
Treatment outcome | 8 to 14 months (2 months after treatment completion)
  Treatment outcomes for patients initiated on treatment according to WHO categories: treatment success, treatment failed, died, lost to follow-up, and not evaluated.
Adherence to the TB treatment | 6 to 12 months (at treatment completion)
  Adherence documented by seven-day recall and counting of pills

CONTACTS AND LOCATIONS:
Overall Officials: Appolinaire Tiam, MBChB, MMed, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (12):
- Cameroon (6):
  - Hopital de District Akonolinga, Akonolinga, Centre Region
  - Hopital de District Soa, Okoa, Centre Region
  - Hopital de District Loum, Loum, Littoral Region
  - Hopital de District Foumban, Mbanga, Littoral Region
  - Hopital de District Dschang, Dschang, West Region
  - Hopital de District Mbouda, Mbouda, West Region
- Kenya (6):
  - Kendu Sub County Hospital, Kendu Bay, Homa Bay County
  - Ndhiwa Sub county Hospital, Ndhiwa, Homa Bay County
  - Kakuma Mission Hospital, Kakuma, Turkana County
  - Lokitaung sub-county hospital, Lokitaung, Turkana County
  - Lopiding Sub County Hospital, Lopiding, Turkana County
  - Homa Bay County Referral Hospital, Homa Bay

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Masaba R, Herrera N, Tchounga B, Siamba S, Ouma M, Okomo G, Tchendjou P, Ditekemena J, Zoung-Kanyi Bissek AC, Casenghi M, Machekano R, Tiam A, Denoeud-Ndam L. Decentralisation and integration of paediatric tuberculosis services to primary healthcare facilities as an approach to optimise management in Cameroon and Kenya: a descriptive cohort study. BMJ Public Health. 2024 Jul 29;2(Suppl 1):e001005. doi: 10.1136/bmjph-2024-001005. eCollection 2024 Jul. PMID 41221323
- [Derived] Tchounga B, Tiam A, Masaba RO, Herrera N, Mbunka M, Siamba S, Goura AP, Ouma M, Petnga SJ, Tchakounte Youngui B, Zemsi A, Zoung-Kanyi Bissek AC, Okomo G, Simo L, Casenghi M, Tchendjou P, Ditekemena J, Rakhmanina N, Denoeud-Ndam L. Assessing tuberculosis clinical presentation, diagnosis and treatment outcomes among children under 5 years old: results from a cohort of children with presumptive TB in Cameroon and Kenya. BMJ Public Health. 2025 Jun 26;2(Suppl 1):e001566. doi: 10.1136/bmjph-2024-001566. eCollection 2024 Jul. PMID 40740312
- [Derived] Katirayi L, Masaba R, Tchounga B, Ndimbii J, Mbunka M, Ouma M, Olughu K, Siehien J, Petnga SJ, Casenghi M, Okomo G, Zoung-Kanyi Bissek AC, Tiam A, Denoeud-Ndam L; INPUT study team. 'We did not even know it was tuberculosis': a qualitative evaluation of integrating tuberculosis services into paediatric entry points in the CaP-TB programme in Cameroon and Kenya. BMJ Public Health. 2024 Jul 2;2(Suppl 1):e001001. doi: 10.1136/bmjph-2024-001001. eCollection 2024 Jul. PMID 40017705
- [Derived] Powell L, Denoeud-Ndam L, Herrera N, Masaba R, Tchounga B, Siamba S, Ouma M, Petnga SJ, Machekano R, Pamen B, Okomo G, Simo L, Casenghi M, Rakhmanina N, Tiam A. HIV matters when diagnosing TB in young children: an ancillary analysis in children enrolled in the INPUT stepped wedge cluster randomized study. BMC Infect Dis. 2023 Apr 17;23(1):234. doi: 10.1186/s12879-023-08216-w. PMID 37069518
- [Derived] Denoeud-Ndam L, Otieno-Masaba R, Tchounga B, Machekano R, Simo L, Mboya JP, Kose J, Tchendjou P, Bissek AZ, Okomo GO, Casenghi M, Cohn J, Tiam A; INPUT Study Group. Integrating pediatric TB services into child healthcare services in Africa: study protocol for the INPUT cluster-randomized stepped wedge trial. BMC Public Health. 2020 May 6;20(1):623. doi: 10.1186/s12889-020-08741-2. PMID 32375741